CLINICAL TRIAL: NCT04647409
Title: Screening for Non-Alcoholic Fatty Liver Disease (NAFLD) in a General Practitioner Population, in Flanders, Belgium.
Brief Title: Screening for NAFLD in Flanders
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Geert Robaeys, Principal Investigator, Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SCREEFLAN-01
Record Dates: First submitted 2020-11-26; First posted 2020-11-30 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participants (Other)
  Interventions: Other: screening

INTERVENTIONS:
Other: screening — The determination of the prevalence of NAFLD in a general population in Flanders, Belgium

SUMMARY:
In the Belgian adult population more than half, and numbers are still increasing, of the population is overweight or obese. These people are at risk to develop NAFLD. However, we lack epidemiological data in Belgium. Therefore, it is important to do epidemiological studies to investigate NAFLD prevalence and disease severity based on a non-invasive approach and evaluate how patients are to be referred.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* able to understand Dutch,
* able to understand the informed consent

Exclusion Criteria:

* secondary causes of steatosis
* excessive alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CLDQ-NAFLD | baseline
  The determination of the prevalence of NAFLD in a general population in Flanders, Belgium by using A disease-specific quality of life instrument for non-alcoholic fatty liver disease and non-alcoholic steatohepatitis
36-Item Short Form Survey (SF-36) | baseline
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and are now widely utilized by managed care organizations and by Medicare for routine monitoring and assessment of care outcomes in adult patients.

CONTACTS AND LOCATIONS:
Overall Officials: Geert Robaeys, prof. dr., Principal Investigator — Hasselt University; Leen Heyens, drs., Study Chair — Hasselt University
Locations (1):
- Hasselt University, Hasselt, Belgium